CLINICAL TRIAL: NCT04743700
Title: "Effects of Piezocision vs Micro-osteoperforations on the Rate of Maxillary Canine Retraction: A Split Mouth Randomized Clinical Trial"
Brief Title: "Effects of Piezocision vs Micro-osteoperforations on the Rate of Maxillary Canine Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Karan.mahendru
Record Dates: First submitted 2020-12-14; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Angle Class II, Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezocision on Experimental Side A (Experimental): Piezocisions with the help of piezotome , mesial and distal to a canine (in a vertical line) with the help of piezotome to accelerate maxillary canine retraction
  Interventions: Procedure: Piezocision
- Micro-osteoperforations on Experimental side B (Experimental): Three MOPs with the help of mini-implant screw driver,mesial and distal to canine(in a vertical line) with the help of minisrew implant driver to accelrate maxillary canine retraction
  Interventions: Procedure: Micro-osteoperforations

INTERVENTIONS:
Procedure: Piezocision — Piezocisions with the help of piezotome , mesial and distal to a canine (in a vertical line) with the help of piezotome. These piezocisions will be performed on the buccal cortical bone only, 2-3mm below the alveolar crest level, 2mm deep into the bone under local anaesthesia (2% lidocaine with 1:100,000 epinephrine) and with standard asepsis, and gingival overlying will be incised first with blade number 15 in a Bard Parker handle . The exact location of incision will be determined by transgingival probing mesial and distal to the canine to know the alveolar crest level and to this measurement 2-3 mm is added and then 5mm incision is given in gingiva and overlying mucoperiosteum in a vertical line apically to expose the underlying bone.
  Arms: Piezocision on Experimental Side A
Procedure: Micro-osteoperforations — Three MOPs mesial and three MOPs distal to canine(in a vertical line) with the help of minisrew implant driver (fig.2). These MOPs will be performed on the buccal cortical bone only, 2-3 mm below the alveolar crest level, 2mm deep into the bone under local anaesthesia (2% lidocaine with 1:100,000 epinephrine) and with standard asepsis, and no flap will be raised. The exact location of first MOP will be determined by transgingival probing mesial and distal to the canine to know the alveolar crest level and to this measurement 2-3 mm is added. The location of second MOP at 5mm apically in a vertical line and third MOP at 5 mm apically to second MOP
  Arms: Micro-osteoperforations on Experimental side B

SUMMARY:
Acceleration of orthodontic tooth movement persuades tremendous rise in the interest of adolescents and aduts, as it not only shortens the treatment duration but also lessens the incidence of white spot lesions, root resorption, periodontal and other soft tissue problems. Minimal invasive techniques i.e.both piezocision and micro-osteoperforations had promising results in accelerating tooth movement. Therefore current study will provide evidence for better minimal invasive technique in terms of reducing treatment time and patient comfort.

DETAILED DESCRIPTION:
Patients with Angle's Class II division 1 malocclusion meeting selection criteria and are indicated for maxillary first premolar extraction, patients will be referred for extraction of the maxillary first premolars , treatment will be initiated by bonding preadjusted MBT 0.022" slot straight wire appliance(Patient will be instructed to report immediately in case of breakage of appliance), after that, leveling and alignment will be done in all subjects, after insertion of 0.019"× 0.025" stainless steel arch wire, alginate impression and periapical radiograph of canine and first molar region will be taken(Before the initiation of canine retraction), randomisation and allocation of two sides of maxillary arch i.e. right and left will be done and active interventions(piezocision and micro-osteoperforations) for each side will be done, immediately maxillary canine retraction will be started with mini-implant and closed NiTi coil spring, patient will be asked to fill pain and discomfort assessment card immediately after initiation of canine retraction., subsequent impressions records will be taken at 4th, 8th, 12th and 16th weeks for measuring rate of maxillary canine retraction, data collection and interpretation of results, further pain assessment cards will be filled after 24 hours, on 7th day and 28th day

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 16-25 years
2. Patients with Angle's class II division 1 malocclusion requiring bilateral extraction of maxillary first premolars.
3. Overjet of ≤ 10mm
4. No debilitating systemic disease.
5. No radiographic evidence of bone loss.
6. No history of periodontal disease/ therapy.
7. No smoking habit.
8. Probing depth of not more than 3mm in all teeth.

Exclusion Criteria:

1. Presence of any signs and symptoms of gingival and periodontal diseases.
2. Overjet more than 10mm.
3. Long-term drug history.
4. Systemic diseases.
5. Evidence of bone loss.
6. Smoking habit.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of rate of canine retraction | 4th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper or acrylic plug method after beginning of maxillary canine retraction
Measurement of rate of canine retraction | 8th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper or acrylic plug method after beginning of maxillary canine retraction
Measurement of rate of canine retraction | 12th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper or acrylic plug method after beginning of maxillary canine retraction
Measurement of rate of canine retraction | 16th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper or acrylic plug method after beginning of maxillary canine retraction

SECONDARY OUTCOMES:
Assessment of pain/discomfort level | at the beginning of canine retraction
  The participants will be asked to assess their level of discomfort on the day of initiation of canine retraction with visual analog scale(VAS).
Assessment of pain/discomfort level | 24 hours
  The participants will be asked to assess their level of discomfort on the day of initiation of canine retraction with visual analog scale(VAS).
Assessment of pain/discomfort level | 7th day
  The participants will be asked to assess their level of discomfort on the day of initiation of canine retraction with visual analog scale(VAS).
Assessment of pain/discomfort level | 28th day
  The participants will be asked to assess their level of discomfort on the day of initiation of canine retraction with visual analog scale(VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No